CLINICAL TRIAL: NCT02033564
Title: Does the Incidence of Sore Throat Increase With the Use of a Traditional Intubation Blade or the Glidescope
Brief Title: Incidence of Sore Throat With Traditional Intubation Blades or Glidescope Blade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jason Ngo, B.S. (Other)
Collaborators: Albany Medical College (Other)
Responsible Party: Sponsor-Investigator, Jason Ngo, B.S., Medical Student, Albany Medical College
Organization: Albany Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3215
Record Dates: First submitted 2014-01-08; First posted 2014-01-13 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Intratracheal Intubation; Laryngoscopes; Postoperative Care; Risk Assessment
Keywords: Sore Throat; Intubation; Laryngoscopy; Anesthesiology; Perioperative; Airway Management
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Macintosh/Miller Laryngoscope (Active Comparator): Macintosh or Miller laryngoscopy blade, preference left up to practitioner conducting intubation. These are the gold standards currently used in laryngoscopy.
  Interventions: Device: Macintosh/Miller Laryngoscope
- Glidescope Laryngoscope (Active Comparator): Glidescope video-guided laryngoscopy blade
  Interventions: Device: Glidescope Laryngoscope

INTERVENTIONS:
Device: Macintosh/Miller Laryngoscope
  Arms: Macintosh/Miller Laryngoscope
Device: Glidescope Laryngoscope
  Arms: Glidescope Laryngoscope

SUMMARY:
The purpose in this study is to determine whether there is a difference in the incidence of postoperative sore throat when using the GlideScope™ versus a traditional intubation blade involving patients that are not anticipated to have a difficult airway.

DETAILED DESCRIPTION:
The goal of this study is to determine whether the use of the GlideScope™ video laryngoscope during intubation leads to a greater or lesser incidence of sore throat when compared to traditional laryngoscope blades used for intubation, such as the Macintosh or Miller blade. During postoperative checks by a board certified anesthesiologist at the Albany Medical Center (AMC) Hospital, it was noticed that patients who reported sore throat often required intubation with the GlideScope™. Standard of care at the AMC Hospital dictates that the Glidescope is used as a "rescue" device for failed direct laryngoscopy on a difficult airway; if traditional direct laryngoscopy with a Macintosh or Miller blade cannot provide adequate laryngeal views, progression to a different airway device such as the Glidescope or fiberoptic scope is indicated. The initial attempt with direct laryngoscopy on a difficult airway often requires utilization of McGill forceps, which increases the chance of upper airway injury prior to the rescue attempt with the GlideScope. Consequently, it is difficult to determine whether patients' reports of post-operative sore throat are caused by the irritation inflicted by the multiple laryngoscopic attempts required in patients where the Glidescope was needed as a rescue method, or whether it is due to the actual utilization of the Glidescope itself.

Previous studies have shown that the use of a GlideScope™ decreases the likelihood of upper airway injury by decreasing the lower mean force applied during laryngoscopy when compared to a Macintosh laryngoscope; however, this study was done using manikins and it is not known whether this result can be translated to a patient oriented outcome. Another study compared the GlideScope™ to direct laryngoscopy for nasotracheal intubation. Their results suggested that the incidence of postoperative moderate or severe sore throat was significantly reduced with use of the GlideScope™ videolaryngoscope. However, other studies have shown increased incidence of postoperative sore throat with Glidescope usage when compared to other videolaryngoscopes and conventional Macintosh laryngoscope as a primary laryngoscopy method. In light of these studies, none have attempted a direct comparison of a Glidescope with conventional Macintosh/Miller laryngoscope blades with incidence of sore throat as a primary outcome of interest.

The purpose in this study is to determine whether there is a difference in the incidence of postoperative sore throat when using the GlideScope™ versus a traditional intubation blade involving patients that are not anticipated to have a difficult airway. Exclusion of patients with difficult airways allows us to perform direct comparisons with the Glidescope and conventional direct laryngoscopy without compromising standard of care or increasing patient risk, which will be determined by the use of standard of care preoperative exams.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 - 80 years old.
* Able to provide written informed consent and to comply with all study procedures
* Scheduled for elective inpatient or outpatient surgery requiring general anesthesia and orotracheal intubation.

Exclusion Criteria:

* Known difficult airway based on prior medical history
* American Society of Anesthesiologists physical status score > IV
* Presence of abnormal cervical spine movement (normal > 90°)
* Airway Mallampati score ≥ III
* Thyromental distance ≥ 6
* Upper lip bite test ≥ 3
* Degree of retrognathia
* Previous medical history indicating patient has a known difficult airway
* Judgment that patient will require intubation post-operatively
* Are emergency surgery cases
* Are Ear-Nose-Throat (ENT) or neck surgery cases
* Have a planned post-operative ICU stay
* Inadequate Nil Per Os (NPO) status prior to surgical case
* Prisoner status

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2012-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Sore Throat | Within 24 hours post-operatively
  Based on subjective yes/no reply by patient

CONTACTS AND LOCATIONS:
Overall Officials: Dennis J Cirilla, DO, Principal Investigator — Department of Anesthesiology, Albany Medical Center
Locations (1):
- Albany Medical Center Hospital, Albany, New York, United States

REFERENCES:
- [Background] Cooper RM, Pacey JA, Bishop MJ, McCluskey SA. Early clinical experience with a new videolaryngoscope (GlideScope) in 728 patients. Can J Anaesth. 2005 Feb;52(2):191-8. doi: 10.1007/BF03027728. PMID 15684262
- [Background] Aziz MF, Healy D, Kheterpal S, Fu RF, Dillman D, Brambrink AM. Routine clinical practice effectiveness of the Glidescope in difficult airway management: an analysis of 2,004 Glidescope intubations, complications, and failures from two institutions. Anesthesiology. 2011 Jan;114(1):34-41. doi: 10.1097/ALN.0b013e3182023eb7. PMID 21150569
- [Background] Carassiti M, Zanzonico R, Cecchini S, Silvestri S, Cataldo R, Agro FE. Force and pressure distribution using Macintosh and GlideScope laryngoscopes in normal and difficult airways: a manikin study. Br J Anaesth. 2012 Jan;108(1):146-51. doi: 10.1093/bja/aer304. Epub 2011 Sep 28. PMID 21965048
- [Background] Jones PM, Armstrong KP, Armstrong PM, Cherry RA, Harle CC, Hoogstra J, Turkstra TP. A comparison of glidescope videolaryngoscopy to direct laryngoscopy for nasotracheal intubation. Anesth Analg. 2008 Jul;107(1):144-8. doi: 10.1213/ane.0b013e31816d15c9. PMID 18635480
- [Background] Teoh WH, Saxena S, Shah MK, Sia AT. Comparison of three videolaryngoscopes: Pentax Airway Scope, C-MAC, Glidescope vs the Macintosh laryngoscope for tracheal intubation. Anaesthesia. 2010 Nov;65(11):1126-32. doi: 10.1111/j.1365-2044.2010.06513.x. Epub 2010 Sep 30. PMID 20883502
- [Background] Higgins PP, Chung F, Mezei G. Postoperative sore throat after ambulatory surgery. Br J Anaesth. 2002 Apr;88(4):582-4. doi: 10.1093/bja/88.4.582. PMID 12066737
- [Background] Dupont WD, Plummer WD Jr. Power and sample size calculations. A review and computer program. Control Clin Trials. 1990 Apr;11(2):116-28. doi: 10.1016/0197-2456(90)90005-m. PMID 2161310
- [Background] Krasser K, Missaghi-Berlini S M, Moser A, Zadrobilek E. Evaluation of the standard adult GlideScope videolaryngoscope: orotracheal intubation performed by novice users after formal instruction. Internet Journal of Airway Management. Available from URL; http://www.ijam.at/volume03/clinicalinvestigation01/default.htm (accessed July 25, 2013).
- [Background] Biro P, Seifert B, Pasch T. Complaints of sore throat after tracheal intubation: a prospective evaluation. Eur J Anaesthesiol. 2005 Apr;22(4):307-11. doi: 10.1017/s0265021505000529. PMID 15892411
- [Background] Sharma D. Is GlideScope the best way to intubate? Anesthesiology. 2010 Jul;113(1):258-9; author reply 259. doi: 10.1097/ALN.0b013e3181e0ef5c. No abstract available. PMID 20574234